CLINICAL TRIAL: NCT02256670
Title: Pilot for The Breast Cancer Endocrine Therapy Adherence (BETA) Trial: Efficacy of a Text-messaging Application in Increasing Adherence With Adjuvant Endocrine Therapy for Stage I-III Hormone Receptor Positive Breast Cancer
Brief Title: Pilot for The Breast Cancer Endocrine Therapy Adherence (BETA) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1409014658
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Hormone Receptor Positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Text Message Application Intervention (Experimental): The study intervention will include a mobile phone two-way text message application. Each prompt described below will generate either a yes (Y)/no (N) or ABCDE(F) response from patients. Each response will generate further prompts resulting in either notification for providers to call patients or relevant phone numbers for patients to call for assistance.
  Interventions: Behavioral: Text Message Application

INTERVENTIONS:
Behavioral: Text Message Application — Two-way text messaging application addressing adherence with adjuvant endocrine therapy
  Other Names: MedAdherence

SUMMARY:
Pilot study to assess feasibility and patient acceptance of a text message cell phone application for patients with stage I-III, hormone receptor positive breast cancer who start adjuvant endocrine therapy.

DETAILED DESCRIPTION:
Approximately 75% of breast cancers express the estrogen and/or progesterone receptor (hormone receptors). The standard of care for women with hormone receptor positive breast cancer is five to ten years of adjuvant endocrine therapy with drugs such as tamoxifen or aromatase inhibitors (AIs). In women with stage I-III breast cancer, treatment with adjuvant endocrine therapy has been shown to reduce recurrences by 30-50% and improve survival. Unfortunately, it is estimated from large population databases that up to 35-40% of patients may discontinue adjuvant endocrine therapy before completing the recommended 5 years for various reasons, and non-adherence may reduce survival.

The current protocol is a pilot study in women with hormone receptor positive breast cancer who are beginning adjuvant endocrine therapy, the purpose of which is to assess the feasibility of a two-way text messaging application, with goals for a larger randomized control study to assess if the application will increase adherence and therefore improve disease free survival. This application includes daily text message medication reminders and periodic assessment of side effects and barriers to medication adherence and simultaneously offers assistance for treatment related issues. The investigators will collect information on QOL and financial burden during the 3 month period and will correlate these metrics with adherence. This larger randomized control study would be the first such interventional study to increase adherence with adjuvant endocrine therapy in breast cancer in the US. Our larger randomized control trial would provide the first longitudinal prospectively collected information on QOL, financial burden and adherence over the entire 5-year treatment period in the routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed stage I-III, estrogen and/or progesterone receptor positive, as defined by ASCO-CAP guidelines, invasive breast cancer for whom adjuvant hormonal therapy is indicated following standard NCCN practice guidelines
* Patients may enter the study before or within one month of starting endocrine treatment
* Patients with synchronous bilateral breast cancers are eligible if both tumors are hormone receptor positive
* Patient must be able to provide informed consent and agree to:
* Complete questionnaires according to the pre-specified study design
* Own a personal cell phone, agree to receive text messages on a monthly basis (including any costs), and share their personal cell phone number to receive text message reminder
* sign consent to allow research staff to contact their pharmacies to determine prescription refill dates

Exclusion Criteria:

* Patients with ductal carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Patient Acceptance of Text Message Program | 3 months
  Using self-report surveys to assess feasibility and patient acceptance of text message program
Adherence to Endocrine Therapy | 3 months
  Adherence rates after 3 months on study, compared with historical controls. Adherence is defined as taking > 80% of prescribed pills based on self reported adherence questionnaire. This threshold was adopted from the literature. Adherence will also be assessed by checking electronic pharmacy dispensation records when feasible.

SECONDARY OUTCOMES:
Quality of Life | 3 months
  Measure quality of life (QOL) and financial burden and correlate with medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mougalian, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States